CLINICAL TRIAL: NCT03710499
Title: Impact of a Physical Rehabilitation Program on the Quality of Life of Patients With Acromegaly: a Non-randomized Clinical Trial.
Brief Title: Rehabilitation Program in Patients With Acromegaly
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centro Universitário Augusto Motta (Other)
Collaborators: Rio de Janeiro State Research Supporting Foundation (FAPERJ) (Other Government); Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Clinical trial in acromegaly
Record Dates: First submitted 2018-10-10; First posted 2018-10-18 (Actual); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Acromegaly; Muscle Dysfunction; Physical Activity; Exercise
Keywords: Acromegaly; Rehabilitation; Physiotherapy
MeSH Terms: conditions — Acromegaly; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: After a physical therapy evaluation, the patient underwent a booklet-guided physical exercise program that lasted two months (3 times per week with a duration of 60 minutes per session). Activities included overall stretching and strengthening (flexion, extension, adduction and abduction movements) and muscular endurance exercises (exercises involving open and closed kinetic chains), along with aerobic conditioning using a functional circuit. The patient was evaluated at 3 different timepoints (baseline, after 8 weeks of training, and after a 4-week washout period with no treatment); thus, he served as his own control. The physiotherapist contacted the patient by phone weekly to follow the progression of the treatment. Throughout the application of the protocol, the patient regularly maintained his follow-up visits with the multidisciplinary team. Moreover, there was no change in pharmacological treatment throughout this period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Physical activity (Experimental): The program comprises the practice of resistance exercises for the main muscular groups, with free weights and with their own body weight against the action of gravity, the proposal consists of 3 weekly sessions, for 8 consecutive weeks.
  Interventions: Procedure: Physical activity

INTERVENTIONS:
Procedure: Physical activity — Activities included overall stretching and strengthening (flexion, extension, adduction and abduction movements) and muscular endurance exercises (exercises involving open and closed kinetic chains), along with aerobic conditioning using a functional circuit.

SUMMARY:
Acromegaly is chronic, systemic and highly disabling disease. People with Acromegaly show a significant reduction in peripheral muscle strength associated with a loss resistance and lethargy. They tend the fatigue more easily when compared to individuals without the disease, which involves exercise intolerance and disability resulting in a quality of life impaired. Acromegaly have important functional limitations that adversely affect the performance in the activities of day-to-day and contribute to the worsening of the disease. Based on previous studies, the investigators believe that acromegaly participants with would have benefit from a treatment protocol facing physical performance and improved quality of life. Main Objective: To evaluate the effect of home rehabilitation on quality of life of participants with acromegaly. Methods: In this study of longitudinal intervention, they will undergo a rehabilitation program lasting three months, three times a week lasting 60 minutes each session. The protocol will be the assessment of Acromegaly Quality of Life Questionnaire (AcroQol) questionnaire, functional assessment by the walk test of six minutes (6MWT), peripheral muscle strength and assessment of joint integrity, fatigue will be measured by the Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) questionnaire that evaluates the fatigue in the chronic participants. The assessment will be in 3 different moment (month 0, month 2 month 3). The treatment protocol will consist of warm-up and cool-down, strengthening exercise and muscular endurance, aerobic training, and balance training and proprioception. Prospects: The participants with acromegaly will benefited significantly after undergoing a physical therapy rehabilitation protocol the following parameters: Resistance and muscle strength, pain conditions and disorders skeletal muscle, improvement in activities of daily living and consequent better quality of life.

DETAILED DESCRIPTION:
Acromegaly is a rare, chronic, disabling disease of endocrine origin that causes several debilitating systemic dysfunctions due to the excessive production of growth hormone (GH) and insulin-like growth factor I (IGF-I) (Gadelha et al., 2017).

In 98% of cases, the disease is caused by a sporadic somatotropinoma. Sporadic somatotropinomas are tumors of monoclonal origin; a mutation that activates the alpha subunit of stimulatory G protein (sgp) is the most common genetic alteration, and it is found in approximately 40% of participants. Somatrotopinomas can be macro- (≥1 cm) or microadenomas (<1 cm); purely GH-secreting (60% of cases), mixed (GH, prolactin, thyroid-stimulating hormone and/or corticotrophin) and occasionally pituitary carcinomas (fewer than 20 published cases); and, even more rarely, hypothalamic neoplasms secreting growth hormone-releasing hormone (GHRH), which stimulates the pituitary gland's production of GH. However, there may occasionally be secondary causes or ectopic sources of GHRH. Typical secondary sources include malignant neoplasms of the adrenals, lungs and pancreas; more rarely, GHRH is secreted by neuroendocrine tumors of the gastrointestinal tract, such as gastrinomas and insulinomas. GH-secreting ectopic tumors (pancreatic islet tumor and non-Hodgkin's lymphoma) occur very rarely (Chanson and Salenave, 2008; Chanson et al., 2009).

In a smaller percentage of cases (5%), the disease may have a familial nature, such as multiple endocrine neoplasia syndromes type 1 and type 4, Carney complex, and familial isolated pituitary adenoma (FIPA), including its subtype, isolated familial somatotropinoma (IFS) (Gadelha et al., 2017; Marques et al., 2017). There are anecdotal reports of the disease being caused by an overdose of GH during treatment for children who do not produce this hormone and in athletes who use GH as a drug to improve muscle performance (Macintyre 1987; Karges et al. 2004).

Chronic exposure to GH and IGF-I has multisystemic repercussions, with changes in metabolic parameters, body composition, cardiac function, pulmonary function, muscle function and exercise capacity, among other effects (Dantas et al., 2013; Hatipoglu et al., 2014; Volschan et al., 2017). IGF-I is produced primarily by the liver (which is responsible for ≈75% of circulating IGF-I) in response to elevated GH levels and, to a lesser extent, to endocrine stimulation of insulin in the liver (Aguirre et al., 2016). Additionally, IGF-I provides an inhibitory feedback signal for GH secretion in the hypothalamus, stimulating the production of somatostatin in the pituitary (Ohlsson et al., 2009). IGF-I is also produced locally in various body tissues, including cartilaginous cells (Aguirre et al., 2016). The availability of IGF-I is tightly regulated by insulin-like growth factor binding proteins (IGFBPs) (Rajpathak et al., 2009). Elevated levels of IGF-I affect several pathways of metabolism, including (1) competition with insulin for the insulin receptor, resulting in diabetes mellitus; (2) general somatic hypertrophy (e.g., macroglossia, acromegalic heart, large kidneys and bulky skeletal muscles); and (3) binding to insulin-like growth factor-1 receptor (IGF-1R), which is a tyrosine kinase receptor that causes the phosphorylation and activation of various intracellular signaling pathways, including the activation of the AKT pathway, which results in the growth and proliferation of somatic cells (Cruzat et al., 2008; Aguirre et al., 2016; Adigun and Mesfin, 2017).

Many of the clinical manifestations of acromegaly are common to other, more prevalent diseases, and diagnosis is often delayed by approximately 8 to 10 years after the onset of the first signs and symptoms (Brue and Castinetti, 2016). Adult participants with acromegaly have the characteristic features of forehead protrusion, nose and lip augmentation, nasolabial sulcus accentuation, prognathism, and enlarged hands and feet (Adigun and Mesfin, 2017). Acromegaly can lead to visceromegaly, hypertension, arrhythmias, cardiomyopathy, diabetes mellitus, ventilatory dysfunction, sleep apnea, osteoarthritis and compressive neuropathies (Colaco et al., 2004; Pivonello et al., 2017). These participants may also present with general fatigue, headache, visual changes, hyperhidrosis, acanthosis nigricans, hypopituitarism, hyperprolactinemia, nephrocalcinosis and an increased incidence of colon and thyroid cancer (Table 1) (Colao et al., 2004). The clinical diagnosis is confirmed biochemically by an elevated IGF-I level for age and a nadir serum GH concentration higher than 1.0 μg/L following an oral glucose tolerance test (Katznelson et al., 2014). The assessment of tumor volume and extent is based on imaging studies using magnetic resonance imaging or computed tomography of the sella turcica (Melmed et al., 2005). The goals of treatment are to correct (or prevent) tumor compression by excision, reduce GH and IGF-I levels to normal, control symptoms, improve quality of life and reduce mortality (Cordido et al., 2013, Leopoldo et al., 2017). Transsphenoidal surgery is the treatment of choice, with exceptions for participants who have a clinical contraindication or who refuse the procedure or in cases of almost entirely unresectable tumors (e.g., those with an epicenter within the cavernous sinus) (Katznelson et al., 2014). When surgery fails to correct GH/IGF-I hypersecretion, adjuvant drug treatment is indicated. At present, there are three classes of drugs available for the treatment of acromegaly: somatostatin receptor ligands, dopaminergic agonists, and GH receptor antagonists (Giustina et al., 2014, Katznelson et al., 2014). Radiation therapy is currently proposed as a third-line treatment (Chanson et al., 2009; Leopoldo et al., 2017). The prognosis of acromegaly has improved in recent years. However, even when participants are cured or their disease is well controlled, sequelae often remain (Leopoldo et al., 2017).

There are innumerable functional limitations that negatively affect the ability of participants with acromegaly to perform activities of daily living (ADLs) and contribute to the deterioration of their health-related quality of life (HRQoL). The dysfunctions that occur in acromegaly mainly involve the bones, joints and muscles, and these structures are affected in almost all cases (Lopes et al., 2014; Lopes et al., 2014; Mazziotti et al., 2018). In participants with acromegaly, progressive damage to the articular and musculoskeletal systems occurs, causing temporomandibular joint dysfunction, hypertrophic arthropathy, chrondrocalcinosis, limitations of joint mobility, genu varum, acroparesthesias, carpal tunnel syndrome, thoracic spine kyphoscoliosis, intermittent claudication (lumbar spinal stenosis) and proximal myopathy (Colao et al., 2004; Chanson and Salenave, 2008; Pivonello et al., 2017). Acromegaly is associated with significant alterations in both peripheral muscle strength and endurance; these participants have reduced muscle strength despite the marked muscular hypertrophy described in previous skeletal muscle biopsy studies (Nagulesparen et al., 1976; Guedes da Silva et al., 2013; Lopes et al., 2015). Acromegalic arthropathy affects both axial and peripheral sites; the knee is the joint most often involved, followed by the shoulder, hip, ankle, elbow and hand joints (Colao et al., 2004; Scacchi and Cavagnini, 2006). Consequently, joint pain had been described in up to 90% of acromegalic participants and negatively impacts their HRQoL (Crespo et al., 2017).

In acromegaly, arthropathy progresses inexorably in advanced stages and unpredictably in smaller ways; it is not influenced by successful treatment of the disease, except in the case of diffuse joint symptoms and some pain sites (Chanson and Salenave, 2008; Chanson et al., 2009). In terms of skeletal muscle, two recent studies showed a paradoxical reduction in muscle mass and an increase in proximal muscle fatigue in participants who achieved biochemical control of acromegaly (Bredella et al., 2017; Füchtbauer et al., 2017). However, to our knowledge, no controlled trial has investigated the effects of successful treatment of the disease on muscle function, as determined by measures of skeletal muscle performance. Given the advances in the treatment of acromegaly, it seems appropriate to assess the impact of these costly interventions on physical performance and functional abilities in participants with different degrees of GH/IGF-I control. Despite the important functional limitations resulting from the involvement of the osteomyoarticular system, rehabilitation programs are currently recommended for this population.

In recent years, HRQoL has been considered as an important factor in the clinical management of acromegaly (Crespo et al., 2017). In these for this patient population, HRQoL is impaired even after clinical treatment and the normalization of the target biochemical values, i.e., GH and IGF-I, which suggests that new therapeutic approaches should be sought to improve functionality (Geraedts et al., 2017, Kyriakakis et al., 2017, Webb et al., 2017). Several investigators have hypothesized the possible benefits of ADL rehabilitation for this group of people, tracing the profile of changes that occur in this population throughout life and identifying the most important points and the main deficiencies and discomforts reported. However, only two studies have objectively evaluated the contributions of regular physical exercise to the physical and cardiovascular performance of acromegalic participants with the aim of characterizing the importance of physical activity in cases of physical and emotional impairments (Hatipoglu et al., 2014; Hatipoglu et al., 2015). Despite these studies, data on physical performance in acromegaly are limited, and physiotherapeutic approaches to such dysfunctions and with their impacts on participants well-being are still poorly established (Dantas et al., 2013, Guedes da Silva et al., 2013, Lopes et al., 2015). The investigators believe that individuals with acromegaly may benefit from a protocol of physiotherapeutic treatment directed towards controlling functional limitations.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acromegaly, of both sexes, older than 18 and younger than 65 years, either with active or controlled disease.
* Patients who present clinical stability and who are eligible for the treatment protocol (patients with hormone deficiency will continue on replacement therapy - SILVA et al., 2013).
* Signature of the Informed Consent Term (TCLE).

Exclusion Criteria:

* Patients with inability to perform the 6MWT, according to ATS criteria.
* Patients who have cognitive impairment by mini mental state examination (MEEN).
* Abandonment of treatment during the application of the protocol.
* Uncontrolled hypertension (> 180/100 mmHg with medication use).
* Use of psychotropic drugs.
* Any significant limitations due to osteoarthropathy.
* History of surgery in the previous year with exercise restriction. Não Untreated hypothyroidism or hypocortisolism (HUBBLE et al., 2014).
* IPAQ with very active classification.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-01-10 (Actual); Primary Completion 2019-09-10 (Estimated); Study Completion 2019-10-10 (Estimated)

PRIMARY OUTCOMES:
Isometric dynamometry with surface electromyography | eight weeks
  Peripheral muscle strength and fatigue strength will be evaluated using an EMG -810 surface electromyograph and a DIN_TRO traction dynamometer. For the strength test, the muscle evaluated will be the femoral quadriceps, the patient will be instructed to perform the knee extension, with the highest possible isometric force. Your positioning will be seated with your hands crossed over the chest, with the upright trunk adjusted by the backrest in order to allow the angle of 90 ° for hip flexion. For analysis of fatigue strength, surface electromyography of the medial vastus muscle (VM) of the dominant lower limb will be used through the 8-channel surface electromyograph from the gross signal. The endurance test consists of a contraction sustained for 60 seconds using 50% of the highest MIVM obtained in the strength test.

SECONDARY OUTCOMES:
Walk test of six minutes (6MWT) | eight weeks
  For the execution of the TC6M, the patient will be previously oriented to use sneakers and comfortable clothing. Later it will be positioned in a corridor of 30 meters, demarcated every 3 meters and oriented to walk as fast as possible, but without running, for a total period of 6 minutes. Peripheral saturation of O2 (SpO2), heart rate (HR), modified Borg scale, blood pressure (BP) during the test will be checked. There will be two tests with a 30 minute interval between them. The distance selected will be the patient's best performance. This is based on reducing the learning effect. Subsequently, the data found will be associated with the forecast of Britto et al. (2013) according to age, height and body weight of each individual.

OTHER OUTCOMES:
Acromegaly Quality of Life Questionnaire (AcroQol) | eight weeks
  The Acromegaly Quality of Life Questionnaire (AcroQol) is a specific, simple and valid instrument for assessing quality of life in people suffering from acromegaly aged 18-70 years. It can be used in two different fields: in clinical trials of new drugs as well as in the follow-up of patients in clinical practice. This is particularly useful in evaluating the effects of intervention or treatment. The questionnaire is one-dimensional and contains 22 items divided into two scales: one that evaluates physical aspects (eight items) and another that evaluates the psychological aspects (14 items). The latter is also divided into two sub-scales: one evaluates physical appearance and another evaluates the impact of the disease on the patient's personal relationships (seven items each). The score is given from 1 to 5 where, the lower the score, the worse the quality of life.
Functional Assessment of Chronic Illness Therapy-Fatigue - (FACIT-F) | eight weeks
  The Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) scale was developed for individuals with chronic diseases to evaluate health-related quality of life, treating fatigue as a multidimensional concept. This scale has been applied in different groups of patients with different types of dysfunctions. FACIT-F is a specific scale of evaluation of fatigue that has good representation of the individual's frame, considered as an instrument of easy application, and its use authorized by the author of the same. It will be answered by the researcher himself, with 13 questions ranging from 0 to 4, where the higher the score, the less fatigue. Your score goes from 0 to 52.
Lower Extremity Functional Scale (LEFS) | eight weeks
  The Lower Extremity Functional Scale (LEFS) is a self-administered questionnaire for orthopedic assessment of lower limb integrity. It was developed according to the concepts of functionality and disability of the World Health Organization (WHO). This scale comprises 20 questions and each has a score that varies between the minimum of zero (extremely difficult) and the maximum of four points (without difficulty). The sum of all items can generate a maximum total of 80 points. Such a level of punctuation suggests a normal functional state, that is, the higher the value obtained, the higher the level of functionality of the individual. The LEFS scale is easy to apply and can be used at different levels of functionality and disability related to the lower limbs. It is usually used in initial evaluations, during treatment and thereafter, in order to establish new therapeutic goals for patients.
Weight (kg) and Height (m) | eight weeks
  Body weight and height of patients will be measured using a Filizola® mechanical scale with a maximum capacity of 150 kilograms and a sensitivity of 100 grams and a stadiometer. Body mass index (BMI) will be calculated by dividing body mass by height squared.
Modified Borg Scale | eight weeks
  Evaluates the perception of the degree of effort, performed during the exercise. Currently, it is used in the modified form described with a score varying with scores between 0 where the level of perception of dyspnea (fatigue) or muscle fatigue is "none" until 10 where the level of perception of dyspnea (fatigue) or muscle fatigue is " maximum".

CONTACTS AND LOCATIONS:
Overall Officials: Tatiana l Lima, Msc, Principal Investigator — Centro Universitário Augusto Motta
Locations (1):
- Centro universitário augusto motta, Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
Data available in scientific environment.